CLINICAL TRIAL: NCT02867800
Title: Abatacept for Graft Versus Host Disease Prophylaxis After Hematopoietic Stem Cell Transplantation for Pediatric Sickle Cell Disease: a Sickle Transplant Alliance for Research Trial
Brief Title: Abatacept for GVHD Prophylaxis After Hematopoietic Stem Cell Transplantation for Pediatric Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Monica Bhatia (Other)
Responsible Party: Sponsor-Investigator, Monica Bhatia, Associate Professor of Pediatrics at the Columbia University Medical Center, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ2350
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease; Graft Versus Host Disease
Keywords: Sickle Cell Disease; Graft Versus Host Disease; Abatacept; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Anemia, Sickle Cell; Graft vs Host Disease | interventions — Diphenhydramine; Acetaminophen; Methylprednisolone; Meperidine; Alemtuzumab; thymoglobulin; fludarabine; fludarabine phosphate; Melphalan; Thiotepa; Cyclosporine; Tacrolimus; Methotrexate; Abatacept; Stem Cell Transplantation; Sirolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Standard GVHD Prophylaxis + Abatacept (Experimental): Subjects will receive
  * premedication (Diphenhydramine, Acetaminophen, Methylprednisolone; and Meperidine as needed)
  * immunosuppression (Alemtuzumab, or Thymoglobulin)
  * conditioning regimen (Fludarabine, Thiotepa, and Melphalan)
  * GVHD prophylaxis: calcineurin inhibitor (Cyclosporine,Tacrolimus, Sirolimus or Mycophenolate Mofetil with permission of the sponsor) and Methotrexate plus Abatacept on days -1, +5, +14 and +28, and a marrow infusion on day 0.
  Interventions: Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Methylprednisolone; Drug: Meperidine; Drug: Alemtuzumab; Drug: Thymoglobulin; Drug: Fludarabine; Drug: Melphalan; Drug: Thiotepa; Drug: Cyclosporine; Drug: Tacrolimus; Drug: Methotrexate; Drug: Abatacept; Procedure: Marrow infusion; Drug: Sirolimus; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Diphenhydramine — (Standard of Care) Premedication
  Diphenhydramine: 1 mg/kg IV or PO q 8 hours (maximum=50 mg)
  Other Names: Benadryl
Drug: Acetaminophen — (Standard of Care) Premedication
  Acetaminophen: 10-15 mg/kg PO q 6 hours (maximum=1000 mg)
  Other Names: Tylenol
Drug: Methylprednisolone — (Standard of Care) Premedication
  Methylprednisolone: 0.25-0.5 mg/kg IV q 6 hours
  Other Names: Medrol
Drug: Meperidine — (Standard of Care) Premedication
  Use as needed (PRN) Meperidine: 0.5 mg/kg IV q 4-6 hours (for rigors)
  Other Names: Demerol
Drug: Alemtuzumab — (Standard of Care) Immunosuppression
  Alemtuzumab:
  A test dose of alemtuzumab, 3 mg, should be administered IV over 2 hours the first day. If the test dose is tolerated, administration of three treatment doses should begin within 24 hours. The three treatment doses should be administered on consecutive days. 10 mg/m2 should be given the first day, 15 mg/m2 the second and 20 mg/m2 the third.
  Other Names: Lemtrada
Drug: Thymoglobulin — (Standard of Care) Immunosuppression
  Thymoglobulin: A 4 mg/kg dose of anti-thymocyte globulin should be administered in place of each alemtuzumab dose not completed.
  Other Names: Genzyme
Drug: Fludarabine — (Standard Conditioning Regimen)
  Fludarabine should be administered 30 mg/m2 IV daily for five days. It should be infused over 30 to 60 minutes.
  Other Names: Fludara
Drug: Melphalan — (Standard Conditioning Regimen)
  Melphalan should be administered 140 mg/m2 IV 3 days before marrow infusion. It should be infused within 60 minutes of preparation and over a maximum of 30 minutes. It should be infused immediately after the fludarabine infusion is complete.
  Other Names: Alkeran
Drug: Thiotepa — (Standard Conditioning Regimen)
  Thiotepa should be administered 8 mg/kg IV 3 days before marrow infusion. It should be infused immediately after the fludarabine infusion is complete. The thiotepa should be infused over one hour.
  Other Names: Thioplex
Drug: Cyclosporine — (Standard GVHD Prophylaxis) Calcineurin inhibitor
  Cyclosporine: Administration will commence no later than at least 36 hours before marrow infusion; Cyclosporine doses will be adjusted to maintain a level of 150-300 ng/ml.
  Other Names: Neoral
Drug: Tacrolimus — (Standard GVHD Prophylaxis) Calcineurin inhibitor
  Tacrolimus: Administration will commence no later than at least 36 hours before marrow infusion; Tacrolimus doses will be adjusted to maintain a level of 8-15 ng/ml.
  Other Names: Protopic
Drug: Methotrexate — (Standard GVHD Prophylaxis)
  Methotrexate will be given at a dose of 15 mg/m2 IV on day 1 and a dose of 10 mg/m2 IV on days 3, 6 and 11. Dosing shall be based on actual weight.
  Other Names: Trexall
Drug: Abatacept — (Investigational)
  Abatacept will be administered intravenously at a dose of 10 mg/kg based on actual weight with a maximum of 750 mg. In cases where the calculated dose is less than or equal to 110% of a simple multiple of a 250 mg vial: 250 mg (275mg), 500 mg (550 mg) or 750 mg (825 mg), the dose may be rounded down to the nearest multiple. No rounding up of the abatacept dose is permitted.
  Other Names: CTLA4-Ig; Orencia
Procedure: Marrow infusion — (Standard)
  A procedure that infuses healthy cells, called stem cells, into your body to replace damaged or diseased bone marrow. A bone marrow transplant may also be used to treat certain types of cancer
  Other Names: stem cell transplant
Drug: Sirolimus — (Standard GVHD Prophylaxis)
  Calcineurin inhibitor (cyclosporine or tacrolimus or with permission of the sponsor: sirolimus or mycophenolate mofetil (MMF)) administration will commence no later than day -2 (at least 36 hours before the stem cell infusion); cyclosporine doses will be adjusted to maintain a level of 150-300 ng/ml. This range assumes monitoring by mass spectrometry. If an immunoassay is used instead, the equivalent range for that immunoassay should be used.
  Other Names: Rapamune
Drug: Mycophenolate Mofetil — (Standard GVHD Prophylaxis)
  Calcineurin inhibitor (cyclosporine or tacrolimus or with permission of the sponsor: sirolimus or mycophenolate mofetil (MMF)) administration will commence no later than day -2 (at least 36 hours before the stem cell infusion); cyclosporine doses will be adjusted to maintain a level of 150-300 ng/ml. This range assumes monitoring by mass spectrometry. If an immunoassay is used instead, the equivalent range for that immunoassay should be used.
  Other Names: MMF

SUMMARY:
To assess the tolerability of the costimulation blocking agent abatacept (CTLA4-Ig) when added to the standard graft versus host disease (GVHD) prophylaxis regimen of a calcineurin inhibitor and methotrexate in patients receiving early alemtuzumab followed by fludarabine, thiotepa, melphalan, and alemtuzumab for conditioning.

DETAILED DESCRIPTION:
Outcomes of hematopoietic stem cell transplantation (HSCT) for children and adolescents with sickle cell disease (SCD) have improved. Graft versus host disease (GVHD), however, remains a barrier to success. GVHD accounts for most of the transplant related mortality and much of the morbidity in this setting-in part through the injury it directly causes and in part through the deleterious effects of steroids and the other immunosuppressive agents used to prevent and treat it. The results of pre-clinical studies and a phase I clinical study in patients with hematologic malignancies suggest that the costimulation blocking agent CTLA4-Ig may hold promise an agent for GVHD prophylaxis. In the present trial, the investigators are assessing the tolerability of adding abatacept to standard GVHD prophylaxis-a calcineurin inhibitor and methotrexate-in pediatric SCD patients receiving early alemtuzumab (completed by day -18) followed by fludarabine, thiotepa, and melphalan for conditioning. This trial will provide the foundation for subsequent trials designed to test the long-term hypothesis that abatacept is a safe, steroid-sparing effective adjunct to standard GVHD prophylaxis in this setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hemoglobin (Hgb) SS or SB0 thalassemia between the ages of 3 and 20.99 years who are at least 10 kg getting an human leukocyte antigen (HLA) matched bone marrow transplant, will be eligible if they are at increased risk for graft versus host disease (GVHD) and have severe SCD.

   (a) Patients falling into one of the following three groups will be considered to be at increased risk for GVHD:

   (i) Are between 10 and 20.99 years and receiving their transplant from an HLA matched related donor.

   (ii) Are between 3 and 9.99 years and receiving their transplant from an HLA matched related donor who is at least 10 years.

   (iii) Are between 3 and 20.99 years and receiving their transplant from an HLA matched unrelated donor. Donors must be matched at the A, B, C and DRB1 loci at the allele level.

   (b) Patients who meet one of the following criteria will qualify as having severe SCD:

   (i) Previous clinical stroke, as evidenced by a neurological deficit lasting longer than 24 hours, which is accompanied by radiographic evidence of ischemic brain injury and cerebral vasculopathy.

   (ii) Asymptomatic cerebrovascular disease, as evidenced by one the following:
   * Progressive silent cerebral infarction, as evidenced by serial MRI scans that demonstrate the development of a succession of lesions (at least two temporally discreet lesions, each measuring at least 3 mm in greatest dimension on the most recent scan) or the enlargement of a single lesion, initially measuring at least 3 mm). Lesions must be visible on T2-weighted MRI sequences.
   * Cerebral arteriopathy, as evidenced by abnormal transcranial doppler (TCD) testing (confirmed elevated velocities in any single vessel of time-averaged maximum mean velocities (TAMMV) > 200 cm/sec for non-imaging TCD) or by significant vasculopathy on magnetic resonance angiogram (MRA) (greater than 50% stenosis of > 2 arterial segments or complete occlusion of any single arterial segment).

   (iii) Frequent ( ≥ 3 per year for preceding 2 years) painful vaso-occlusive episodes (defined as episode lasting ≥ 4 hours and requiring hospitalization or outpatient treatment with parenteral opioids). If patient is on hydroxurea and its use has been associated with a decrease in the frequency of episodes, the frequency should be gauged from the 2 years prior to the start of this drug.

   (iv) Recurrent ( ≥ 3 in lifetime) acute chest syndrome events which have necessitated erythrocyte transfusion therapy.

   (v) Any combination of ≥ 3 acute chest syndrome episodes and vaso-occlusive pain episodes (defined as above) yearly for 3 years. If patient is on hydroxurea and its use has been associated with a decrease in the frequency of episodes, the frequency should be gauged from the 3 years prior to the start of this drug.
2. All patients and/or their parents or legal guardians must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
3. Must have been evaluated and adequately counseled regarding treatment options for severe SCD by a pediatric hematologist.
4. Because of the elective and non-urgent nature of hematopoietic stem cell transplantation (HSCT) for SCD, it is important that all patients and families be counseled regarding fertility preservation measures available to them. All patients and/or their parents or legal guardians must indicate on the consent and assent forms that they have received this counseling.

Exclusion Criteria:

1. Bridging (portal to portal) fibrosis or cirrhosis of the liver.
2. Parenchymal lung disease stemming from SCD or other process defined as a diffusing capacity of the lungs for carbon monoxide (DLCO) (corrected for hemoglobin) or forced vital capacity of less than 45% of predicted. Children unable to perform pulmonary function testing will be excluded if they require daytime oxygen supplementation.
3. Renal dysfunction with an estimated glomerular filtration rate (GFR) < 50% of predicted normal for age.
4. Cardiac dysfunction with shortening fraction < 25%.
5. Neurologic impairment other than hemiplegia, defined as full-scale IQ ≤70, quadriplegia or paraplegia, inability to ambulate, or any impairment resulting in decline of Lansky performance score to < 70%.
6. Clinical stroke within 6 months of anticipated transplant.
7. Karnofsky or Lansky functional performance score < 70%.
8. Patient is human immunodeficiency virus (HIV) infected.
9. Donor is HIV infected.
10. Donor has Hgb SS, SC or SB0 thalassemia.
11. Patient with unspecified chronic toxicity serious enough to detrimentally affect the patient's capacity to tolerate bone marrow transplantation.
12. Patient or patient's guardian(s) unable to understand the nature and risks inherent in the bone marrow transplant (BMT) process.
13. History of lack of compliance with medical care that would jeopardize transplant course.
14. Donor who for psychological, physiologic, or medical reasons is unable to tolerate a bone marrow harvest or receive general anesthesia.
15. Active viral, bacterial, fungal or protozoal infection.
16. Donor is pregnant.
17. Patient is pregnant.

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Number of patients who tolerate abatacept | Within 100 days of receiving the last prescribed dose of abatacept
  Patients will be deemed to be evaluable for tolerability if they received all prescribed doses of abatacept.
  Abatacept will deemed to be tolerated, if no more than one dose is withheld per protocol stipulations, no death from an infection that occurs within 30 days of or develops post-transplant lymphoproliferative disease (PTLD) within 100 days of receiving the last prescribed dose of abatacept.

SECONDARY OUTCOMES:
Bearman Scale Score of Regimen-Related Toxicity (RRT) | Day 42 post-transplant
  RRT will be assessed according to Bearman Scale.
Number of infections | Up to 180 days post transplant
  Infections will include viremia, posttransplant lymphoproliferative disease and immune reconstitution.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Bhatia, MD, Study Chair — Columbia University
Locations (7):
- United States (7):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - North Carolina Cancer Hospital, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No